CLINICAL TRIAL: NCT03140722
Title: Phase 2, Randomized, Open-Label Study Evaluating the Efficacy and Safety of Oral Vadadustat for the Treatment of Anemia in Subjects With Dialysis-Dependent Chronic Kidney Disease (DD-CKD) Who Are Hyporesponsive to Erythropoiesis Stimulating Agents
Brief Title: Study to Evaluate Vadadustat for Anemia in Subjects With Dialysis-Dependent Chronic Kidney Disease (DD-CKD) Who Are Hyporesponsive to Erythropoiesis Stimulating Agents
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Revised study design.
Sponsor: Akebia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AKB-6548-CI-0018
Record Dates: First submitted 2017-05-03; First posted 2017-05-04 (Actual); Results first posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Anemia; Dialysis-Dependent Chronic Kidney Disease
Keywords: anemia; kidney; dialysis-dependent chronic kidney disease; CKD; DD-CKD; renal; vadadustat; AKB-6548; hypoxia-inducible factor; HIF; hypoxia-inducible factor prolyl-hydroxylase inhibitor; HIF-PHI; hyporesponder; hyporesponsive; epoetin alfa; hemoglobin; erythropoiesis stimulating agent; ESA
MeSH Terms: conditions — Anemia | interventions — vadadustat; Epoetin Alfa

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- vadadustat (Experimental): Vadadustat daily oral dose, adjustable based on Hb level
  Interventions: Drug: vadadustat
- epoetin alfa (Active Comparator): Epoetin alfa, dose adjustable based on Hb level, as clinically indicated throughout the study
  Interventions: Drug: epoetin alfa

INTERVENTIONS:
Drug: vadadustat — vadadustat
  Other Names: AKB-6548
  Arms: vadadustat
Drug: epoetin alfa — epoetin alfa
  Arms: epoetin alfa

SUMMARY:
This is a Phase 2, randomized, open-label study to evaluate vadadustat versus epoetin alfa for the treatment of anemia in subjects with Dialysis-dependent Chronic Kidney Disease (DD-CKD) who are hyporesponsive to erythropoiesis stimulating agents (ESAs.)

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥18 years of age
* Receiving chronic maintenance hemodialysis for end-stage kidney disease
* Currently receiving epoetin alfa for anemia
* Hb between 8.5 and 10.0 g/dL during screening

Exclusion Criteria:

* Anemia due to a cause other than CKD or presence of active bleeding or recent blood loss
* Sickle cell disease, myelodysplastic syndromes, bone marrow fibrosis, hematologic malignancy, myeloma, hemolytic anemia, thalassemia, or pure red cell aplasia
* Red blood cell transfusion within 4 weeks prior to or during screening
* Anticipated to recover adequate kidney function to no longer require hemodialysis during study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-03-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Akebia Therapeutics, Study Director — Sponsor GmbH
Locations (18):
- United States (18):
  - Research Site, Bakersfield, California
  - Research Site, Elk Grove, California
  - Research Site, Encino, California
  - Research Site, Escondido, California
  - Research Site, Lynwood, California
  - Research Site, San Diego, California
  - Research Site, San Luis Obispo, California
  - Research Site, Waterbury, Connecticut
  - Research Site, Miami, Florida
  - Research Site, Orlando, Florida
  - Research Site, Statesboro, Georgia
  - Research Site, Detroit, Michigan
  - Research Site, The Bronx, New York
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, El Paso, Texas
  - Research Site, Houston, Texas
  - Research Site, Newport News, Virginia
  - Research Site, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Vadadustat: Participants were to discontinue epoetin alfa, administered during the 28-day Screening Period, and initiate vadadustat on Day 1 of the 20-week treatment period. The vadadustat daily oral dose was adjustable based on the target hemoglobin (Hb) level of 10.0 to 11.0 grams per deciliter (g/dL).
- Epoetin Alfa: Participants were to receive the same dose of epoetin alfa administered during the 28-day Screening Period starting on Day 1 of the 20-week Treatment Period. Epoetin alfa was administered based on the approved label for adult participants with Chronic Kidney Disease (CKD) on dialysis, and the dose was adjustable based on Hb level, as clinically indicated throughout the study.
Period: Overall Study
Arm/Group | Vadadustat | Epoetin Alfa
Started | 0 | 2
Completed | 0 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All subjects enrolled in the trial.
Groups:
- Total: Total of all reporting groups
Arm/Group | Vadadustat | Epoetin Alfa | Total
Number analyzed (Participants) | 0 | 2 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years |  | 0 | 0
  Between 18 and 65 years |  | 1 | 1
  >=65 years |  | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Asian |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Native Hawaiian or Other Pacific Islander |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Black or African American |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.
  White |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.
  More than one race |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.
  Unknown or Not Reported |  | NA — Reporting demographic data for this study in which only 2 participants were enrolled introduces the risk of participant identification. In order to protect the participant's privacy, results for the study cannot be reported. | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Hemoglobin (Hb) Over Time During the Treatment Period
Time Frame: Baseline; up to 20 weeks
Population: No efficacy analyses were conducted due to the limited number of participants enrolled prior to study termination (N=2). In order to protect the privacy of participants, the results of enrolled participants cannot be reported.
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Number of Participants Demonstrating Incremental Increases in Hb From Baseline Over Time During the Treatment Period
Time Frame: Baseline; up to 20 weeks
Population: as for outcome 1
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Participants With Hb Values Within the Target Range of 10.0-11.0 Grams Per Deciliter (g/dL) During the Treatment Period
Time Frame: Baseline; up to 20 weeks
Population: as for outcome 1
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Participants Receiving Epoetin Alfa Rescue
Time Frame: up to 20 weeks
Population: as for outcome 1
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Number of Participants Receiving Red Blood Cell Transfusion
Time Frame: up to 20 weeks
Population: as for outcome 1
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Participants With Specified Levels of Various Biomarkers, Including C-reactive Protein, Hepcidin, and Vascular Endothelial Growth Factor
Time Frame: up to 20 weeks
Population: as for outcome 1
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Mean Weekly Dose of Intravenous Elemental Iron Administered
Time Frame: up to 20 weeks
Population: as for outcome 1
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Number of Participants Maintaining Iron Sufficiency (Defined as Ferritin ≥100 Nanograms Per Milliliter and Transferrin Saturation ≥20%)
Time Frame: up to 20 weeks
Population: as for outcome 1
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Number of Participants Utilizing Resources
Time Frame: up to 20 weeks
Population: as for outcome 1
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Treatment-emergent adverse events were collected in all participants enrolled in the study.
Time Frame: up to 24 weeks
Population: All participants enrolled in the study
Measure: Count of Participants; unit: Participants
Arm/Group | Vadadustat | Epoetin Alfa
Number analyzed (Participants) | 0 | 2
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: up to Week 24
Description: No participants were enrolled in the vadadustat arm of the study.
Arm/Group | Vadadustat | Epoetin Alfa
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

LIMITATIONS AND CAVEATS:
The Study was closed by the Sponsor as it was determined that it was more appropriate to initiate a new study that would explore the broader population utilizing a modified dosing approach (rather than amending the current protocol design).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-18): https://cdn.clinicaltrials.gov/large-docs/22/NCT03140722/Prot_SAP_000.pdf